CLINICAL TRIAL: NCT06584643
Title: Evaluation of Serum Gasdermin D Level As a Potential Biomarker of Disease Activity in Vitiligo Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ashraf Sayed Abdelghany, doctor, Assiut University
Other Study IDs: Serum Gasdermin D in vitiligo
Record Dates: First submitted 2023-12-18; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-11

CONDITIONS: Serum Gasdermin D in Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case group: For every patient, a full history will be taken recording age, gender, education, residence, special habits, age at onset of vitiligo, duration of vitiligo, stability of vitiligo and family history. A detailed cutaneous examination will be performed including skin phototype, Koebner phenomenon, vitiligo clinical type, leukotrichia, Vitiligo Area Severity Index (VASI) and Vitiligo Disease Activity (VIDA) scores.
  Interventions: Diagnostic Test: gasdermin d
- healthy control: age and gender matched healthy volunteers as controls
  Interventions: Diagnostic Test: gasdermin d

INTERVENTIONS:
Diagnostic Test: gasdermin d — evaluation of serum gasdermin d in vitligo patients and healthy controls

SUMMARY:
Assessment the serum level of Gasdermin D level in vitiligo patients. Correlate its level with disease activity scores using Vitiligo Area Severity Index (VASI) and Vitiligo Disease Activity (VIDA) scores and with different disease parameters.

DETAILED DESCRIPTION:
Vitiligo, a common depigmenting skin disorder, has an estimated prevalence of 0.5-2% of the population worldwide. The disease is characterized by the selective loss of melanocytes which results in typical nonscaly, chalky-white macules. In recent years, considerable progress has been made in our understanding of the pathogenesis of vitiligo which is now clearly classified as an autoimmune disease .

The destruction of melanocyte is thought to be of multifactorial causation. Genome-wide associated studies have identified single-nucleotide polymorphisms in a panel of susceptible loci as risk factors in melanocyte death. But vitiligo onset can't be solely attributed to a susceptive genetic background .

Oxidative stress triggered by elevated levels of reactive oxygen species accounts for melanocytic molecular and organelle dysfunction, in addition to the self-responsive immune function directly contributes to the bulk of melanocyte deaths in vitiligo .

Moreover, apoptosis is the most extensively documented way of melanocyte demise, with few melanocytes undergo necrosis. But forms of cell death are not merely restricted to apoptosis and necrosis. Cells may die from accidental cell death (ACD) or regulated cell death (RCD). ACD, like necrosis, is biologically uncontrolled, whereas RCD (apoptosis, necroptosis, pyroptosis, oxeiptosis, ferroptosis, parthanatos, etc.) involves precise signaling cascade and molecular mechanisms .

Pyroptosis is mechanistically distinct from other forms of cell death with gasdermin D (GSDMD) and caspase-1/4/5/11 activation as its defining feature . Upon being stimulated by damage-associated molecular patterns molecules (DAMPs), pathogen-associated molecular patterns molecules or altered homeostasis, caspases are activated to cleave the downstream GSDMD. GSDMD fragment with membrane pore-forming activity yields plasma membrane rupture, cytosolic content release, and concurrent cell swelling and lysis

Gasdermins belong to the pore-forming protein family and consist of six gasdermin proteins, including gasdermins A-E. The members of the gasdermin family have two domains: an N-terminal domain and a C-terminal domain linked by a flexible peptide. Upon activation, the cleaved N-terminal domain is responsible for inducing pyroptosis . GSDMD, the most extensively studied executive pyroptosis-executing protein with the clearest mechanism.

In a previous study, scRNA-seq datasets of skin-derived cells from healthy donors and patients with vitiligo were analysed. Results demonstrated that CASP1, CASP4, CASP6, CASP8, and GSDMD expression was significantly upregulated in melanocytes of patients with vitiligo. These results indicated that pyroptosis signaling is an important pathway in the development of vitiligo .

To the best of our knowledge, no previous studies have evaluated the serum level of Gasdermin D as a potential biomarker in vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* All clinically diagnosed cases of vitiligo (segmental and non-segmental).

Exclusion Criteria:

1. patients with inflammatory diseases.
2. patients with autoimmne diseases.
3. patients with neurodegenerative diseases.
4. patients with HIV or COVID19 infection or any other type of infections.
5. patients with systemic diseases as liver diseases or having tumors.
6. patients who received systemic treatment in the last 3 months or topical treatment 1 month prior to the study.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For every patient, a full history will be taken recording age, gender, education, residence, special habits, age at onset of vitiligo, duration of vitiligo, stability of vitiligo and family history. A detailed cutaneous examination will be performed including skin phototype, Koebner phenomenon, vitiligo clinical type, leukotrichia, Vitiligo Area Severity Index (VASI) and Vitiligo Disease Activity (VIDA) scores.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment the serum level of Gasdermin D level in vitiligo patients | basline
  estimate the serum level of Gasdermin D level in vitiligo patients and correlate its level with disease activity and various disease parameters.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergqvist C, Ezzedine K. Vitiligo: A Review. Dermatology. 2020;236(6):571-592. doi: 10.1159/000506103. Epub 2020 Mar 10. PMID 32155629
- [Background] Chen J, Li S, Li C. Mechanisms of melanocyte death in vitiligo. Med Res Rev. 2021 Mar;41(2):1138-1166. doi: 10.1002/med.21754. Epub 2020 Nov 17. PMID 33200838
- [Background] Shi J, Gao W, Shao F. Pyroptosis: Gasdermin-Mediated Programmed Necrotic Cell Death. Trends Biochem Sci. 2017 Apr;42(4):245-254. doi: 10.1016/j.tibs.2016.10.004. Epub 2016 Dec 5. PMID 27932073
- [Background] Broz P, Pelegrin P, Shao F. The gasdermins, a protein family executing cell death and inflammation. Nat Rev Immunol. 2020 Mar;20(3):143-157. doi: 10.1038/s41577-019-0228-2. Epub 2019 Nov 5. PMID 31690840
- [Background] Shi J, Zhao Y, Wang K, Shi X, Wang Y, Huang H, Zhuang Y, Cai T, Wang F, Shao F. Cleavage of GSDMD by inflammatory caspases determines pyroptotic cell death. Nature. 2015 Oct 29;526(7575):660-5. doi: 10.1038/nature15514. Epub 2015 Sep 16. PMID 26375003
- [Background] Rogers C, Fernandes-Alnemri T, Mayes L, Alnemri D, Cingolani G, Alnemri ES. Cleavage of DFNA5 by caspase-3 during apoptosis mediates progression to secondary necrotic/pyroptotic cell death. Nat Commun. 2017 Jan 3;8:14128. doi: 10.1038/ncomms14128. PMID 28045099
- [Background] Zhang D, Li Y, Du C, Sang L, Liu L, Li Y, Wang F, Fan W, Tang P, Zhang S, Chen D, Wang Y, Wang X, Xie X, Jiang Z, Song Y, Guo R. Evidence of pyroptosis and ferroptosis extensively involved in autoimmune diseases at the single-cell transcriptome level. J Transl Med. 2022 Aug 12;20(1):363. doi: 10.1186/s12967-022-03566-6. PMID 35962439
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] Rossiter ND, Chapman P, Haywood IA. How big is a hand? Burns. 1996 May;22(3):230-1. doi: 10.1016/0305-4179(95)00118-2. PMID 8726264
- [Background] Kawakami T, Hashimoto T. Disease severity indexes and treatment evaluation criteria in vitiligo. Dermatol Res Pract. 2011;2011:750342. doi: 10.1155/2011/750342. Epub 2011 May 22. PMID 21747840
- [Background] Njoo MD, Das PK, Bos JD, Westerhof W. Association of the Kobner phenomenon with disease activity and therapeutic responsiveness in vitiligo vulgaris. Arch Dermatol. 1999 Apr;135(4):407-13. doi: 10.1001/archderm.135.4.407. PMID 10206047